CLINICAL TRIAL: NCT05095272
Title: Induced Blood-Stage Plasmodium Vivax Infection With HMPBS02-Pv Challenge Agent in Healthy Malaria-Naive Adults to Produce a Plasmodium Vivax Parasite Cell Bank for Future Studies
Brief Title: Blood-Stage Plasmodium Vivax Cell Bank
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10000212; 000212-I
Record Dates: First submitted 2021-10-26; First posted 2021-10-27 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-08

CONDITIONS: Malaria
Keywords: Malaria; Parasitemia; IBSM; inoculation; Challenge
MeSH Terms: conditions — Malaria; Parasitemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy malaria-naive US adults (Experimental): A single dose of cryopreserved inoculum containing blood-stage P. vivax will be administered IV
  Interventions: Biological: HMPBS02-Pv

INTERVENTIONS:
Biological: HMPBS02-Pv — The blood-stage P. vivax master cell bank HMPBS02-Pv was also produced using blood collected from a consenting patient with naturally acquired malaria infection. The malaria infection was confirmed to be P. vivax by species-specific PCR at Pathology Queensland (accredited by the Australian National Association of Testing Authorities) and further confirmed by deep sequencing at the Sanger Institute. The clinical response to antimalarial chemotherapy was also demonstrated with this donor, who was successfully cured with artemether/lumefantrine.

SUMMARY:
Background:

Malaria is caused by a parasite (a type of germ called P. vivax) that is carried by mosquitoes. The disease is transmitted to people when they are bitten by infected mosquitoes. To make drugs and vaccines for malaria, researchers need malaria-infected blood. Plasmodium vivax cell cultures are currently not cultured in vivo, and thus establishing a blood bank from P. vivax infections will be vital for future research.

Objective:

The goal of this study is to infect people with early-stage malaria, then collect infected blood samples to store in a cell bank for future use.

Eligibility:

Healthy adults ages 18-50 who will not be living alone during the study period.

Design:

Participants will be screened with a physical exam, heart health test, and medical history. They will have blood and urine tests. They will take a mental health survey. They must pass an exam to prove they understand the study.

Participants will have red blood cells infected with P. vivax injected into an arm vein. They will be observed for side effects. They will get a thermometer to measure their temperature at home.

For the next 3 days, they will be monitored via phone call or text. Starting on day 4 after the infection, they will have daily study visits to give blood samples. They will likely develop symptoms of malaria, such as fever, chills, headache, and muscle pain.

Participants will be admitted to the hospital for 2-3 days when either they develop symptoms or the daily blood tests detect a certain amount of parasites. Once malaria is confirmed, a sample of their blood will be collected for the cell bank. Then they will be treated for malaria with oral medication that will cure the infection. Those who do not develop malaria will begin treatment after 15 days.

Participants will have follow-up visits 28 and 90 days after infection.

Participation will last for 3-5 months.

DETAILED DESCRIPTION:
This is a single-center, open-label study using induced blood-stage malaria (IBSM) to produce a human malaria parasite (HMP) bank for use in future studies. This study will be conducted in up to two participants. Participants will be inoculated intravenously (IV) with human malaria parasite blood stage P. vivax (HMPBS02-Pv) parasite-infected erythrocytes (day 0) and then monitored closely via outpatient clinic visits, phone visits, and while inpatient at the NIH Clinical Center (CC) for symptoms and signs of malaria to characterize the safety, tolerability, and infectivity in healthy malaria-naive participants inoculated with P. vivax. Blood sampling will be done periodically to measure parasitemia via quantitative polymerase chain reaction (qPCR) targeting the P. vivax 18S rRNA gene.

The threshold for the commencement of collection of blood for production of the HMP bank and subsequent antimalarial rescue treatment with artemether/lumefantrine will occur when the Malaria Clinical Score is >6 (admission within 24 hours of notification), or parasitemia is >20,000 parasites/mL, or at the investigator s discretion. When this threshold is reached, the participant will be admitted to the NIH CC for further safety assessments before undergoing the blood collection procedure.

After blood collection, the first dose of artemether/lumefantrine will be administered and the participant will remain inpatient for 48-72 hours to monitor for safety and tolerability of rescue therapy, and to ensure adequate clinical and parasitological response to treatment. In the unlikely and unprecedented event that artemether/lumefantrine fails to clear parasitemia, participants will be treated with chloroquine. If oral administration of either artemether/lumefantrine or chloroquine is not possible (e.g., the participant is vomiting), the participant will receive IV treatment with artesunate. After discharge, participants will be followed on an outpatient basis for monitoring of safety and parasite clearance. Follow-up for safety assessments will be performed on day 28 plus or minus 3, day 56 plus or minus 7 (phone call only), and day 90 plus or minus 7 (End of Study).

Participants may also be evaluated for the presence of sexual parasite stages (gametocytes) and other parasite lifecycle stages in the blood during the study using quantitative reverse transcriptase PCR (qRT-PCR).

Objectives: Primary Objective: The collection of blood from healthy participants experimentally infected with P. vivax isolate HMPBS02-Pv for the production of a P. vivax blood-stage parasite bank for use in future studies.

Secondary Objective: To assess the safety and tolerability of the P.vivax IBSM model following inoculation of healthy malaria-naive participants with P. vivax.

Exploratory Objective: To further characterize blood- and sexual stage parasite growth profiles following inoculation with P. vivax isolate and treatment with artemether/lumefantrine.

Endpoints: Primary Endpoint: Collection of blood for the production of a P.vivax blood-stage parasite bank from study participants following experimental infection with P. vivax isolate HMPBS02-Pv.

Secondary Endpoint: Occurrence of solicited and unsolicited adverse events (AEs) following P. vivax inoculation prior to the initiation of antimalarial treatment.

Exploratory Endpoint: The rate of growth of blood- and sexual-stage P. vivax isolate following inoculation and treatment with artemether/lumefantrine as determined by blood smear and/or qPCR.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a participant to participate in this trial:

* Age >=18 and <=50 years.
* In good general health and without clinically significant medical history.
* Does not live alone from study Day 0 until the end of the antimalarial drug treatment.
* Malaria comprehension exam completed, passed (a score of >=80% or per investigator s discretion) and reviewed prior to enrollment.
* Reliable access to the NIH CC and availability to participate for duration of study.
* Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to study Day 0 to 28 days following IBSM.
* Sign written informed consent prior to undertaking any study-related procedure.

EXCLUSION CRITERIA:

A participant will be excluded from participating in this trial if any one of the following criteria is fulfilled:

* Currently breastfeeding (if female).
* Pregnant as determined by a positive urine or serum human choriogonadotropin (Beta-hCG) test (if female).
* Planned travel to a malaria-endemic area during the study period and up to 2 weeks following the EOS visit.
* History of recent travel to or residence in a P. vivax malaria-endemic region for more than 2 weeks during the past 5 years.
* Planned travel to a malaria-endemic region during the course of the study (for endemic regions, see www.cdc.gov/malaria/travelers/country_table).
* Any history of confirmed malaria diagnosis on peripheral blood smear or by clinical history
* Participation in a previous malaria challenge study.
* Screening laboratory parameters outside of local lab normal range, to include serum-corrected calcium, creatinine, hepatic transaminase enzymes (ALT, AST), total bilirubin (unless the participant has documented Gilbert syndrome), and hemoglobin. Participants may be included at the investigator s discretion for not clinically significant values outside of normal range.
* Abnormal urinalysis as defined by positive urine glucose, protein, and hemoglobin. Participant can be included if investigator determine the abnormality is not clinically significant.
* Duffy blood group negative (male or female).
* ABO blood type other than O (male or female).
* Rh blood group negative (females of childbearing potential).
* Anticipated use during the study period, or use within the following periods prior to enrollment of any of the following: Investigational malaria vaccine within the last 2 years; Malaria chemoprophylaxis within the past 6 months; Chronic systemic immunosuppressive medications (>14 days) within 6 months; Blood products or immunoglobulins within the previous 6 months; Systemic antibiotics or medications with potential antimalarial effects within the past 6 weeks; Investigational or non-registered product or vaccine within 30 days; Receipt of any vaccination within 28 days prior to P. vivax IBSM; Medications known to interact with artemether/lumefantrine; Anticoagulants within the past 28 days.
* History of:

  * Sickle cell disease, sickle cell trait, or other hemoglobinopathies.
  * Splenectomy or functional asplenia.
  * Systemic anaphylaxis.
  * Any allergic reactions to artemether/lumefantrine, chloroquine (or any 4-aminoquinolines), artemether or other artemisinin derivatives, or their excipients.
  * History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.
  * Blood transfusion.
* Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status and participation in the study in the opinion of the investigator.
* Vital signs taken after 5 minutes of resting in seated or supine position that fall outside the following ranges:

  * Systolic blood pressure <=90 mm Hg or >=140 mm Hg.
  * Diastolic blood pressure <=50 mm Hg or >=90 mm Hg.
  * Heart rate <=40 bpm or >=100 bpm.
* Body mass index less than 17.0 or greater than 35.0 kg/m2 at the time of screening.
* History of, or known active cardiac disease including: (1) prior myocardial infarction (heart attack); (2) angina pectoris; (3) congestive heart failure; (4) valvular heart disease; (5) cardiomyopathy; (6) pericarditis; (7) stroke or transient ischemic attack; (8) exertional chest pain or shortness of breath; (9) symptomatic cardiac arrhythmias; (10) clinically relevant bradycardia; or (11) other heart conditions under the care of a doctor.
* Clinically significant electrocardiogram (ECG) findings as determined by the expert study cardiologist, or QTcF >=450 ms, or presence of second- or third-degree atrioventricular block or abnormal T wave morphology.
* Moderate or high risk for coronary heart disease based on National Health and Nutrition Examination Survey (NHANES) I cardiovascular risk assessment (Appendix A).
* Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
* History of electrolyte disturbances, particularly hypokalemia, hypocalcemia, or hypomagnesemia.
* Acute infectious disease or fever (e.g., temperature >=38.5 degrees C) within the 5 days prior to inoculation with malaria parasites.
* Evidence of acute illness within the 4 weeks prior to screening that the investigator deems may compromise participant safety.
* Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) antibodies, and anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive urine drug test for any drug unless there is an explanation acceptable to the investigator.
* Elevated serum ethanol level.
* Psychiatric condition that precludes compliance with the protocol.
* Suspected or known current alcohol or drug abuse as defined by the American Psychiatric Association in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, at the discretion of the investigator.
* Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking for the duration of admission. Participants may smoke up to 5 cigarettes or equivalent per day for the rest of the study.
* History or presence of alcohol abuse (alcohol consumption of more than 4 standard drinks per day), drug habituation, or any prior intravenous usage of an illicit substance.
* Excessive consumption of beverages or food containing xanthine bases (such as Red Bull, chocolate, etc.), or more than 400 mg of caffeine per day (equivalent to more than 4 cups of coffee per day).
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will be advised by phone not to consume any poppy seeds in this time period).
* Use of prescription drugs or non-prescription drugs and herbal supplements (such as St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the inoculation administration. (Note: diazepam interferes with the analysis of blood levels of chloroquine and thus should not have been used for at least 8 weeks prior to administration of the study drug). If needed (i.e., an incidental and limited need), ibuprofen up to 1.2 g/day or acetaminophen up to 4 g/day is acceptable. The participant must inform the investigator of any ibuprofen or acetaminophen use at the next convenient time. Limited use of other non-prescription medications or dietary supplements not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor in consultation with the investigator. Participants are requested to refrain from taking non-approved concomitant medications from recruitment until the conclusion of the study.
* Clinical trial staff with direct involvement in the conduct of the trial are excluded from participation.
* Participating in other clinical trials involving investigational interventions or off-label medication use during the study period or within the 12 weeks preceding study day 0. Participation in other trials such as observational or imaging studies will be discussed with the investigators.
* Blood donation of any volume within 4 weeks prior to study day 0, or participation in any research study involving blood sampling (more than 450 mL/unit of blood), or blood donation to Red Cross (or other) blood bank within 8 weeks prior to study day 0.
* Unwillingness to defer blood donations for at least 3 years.
* Unwillingness to abstain from consumption of quinine-containing foods/beverages, such as tonic water or lemon bitter, from inoculation (study day 0) to the end of antimalarial treatment.
* Unwillingness to abstain from consumption of grapefruit or Seville oranges from inoculation (study day 0) to the end of antimalarial treatment.
* Any participant without a good peripheral venous access.
* Participant who, in the judgment of the investigator, is likely to be noncompliant during the study, or is unable to cooperate because of a language or mental deficit.
* Any other finding that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant s ability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffin P, Pasay C, Elliott S, Sekuloski S, Sikulu M, Hugo L, Khoury D, Cromer D, Davenport M, Sattabongkot J, Ivinson K, Ockenhouse C, McCarthy J. Safety and Reproducibility of a Clinical Trial System Using Induced Blood Stage Plasmodium vivax Infection and Its Potential as a Model to Evaluate Malaria Transmission. PLoS Negl Trop Dis. 2016 Dec 8;10(12):e0005139. doi: 10.1371/journal.pntd.0005139. eCollection 2016 Dec. PMID 27930652
- [Background] McCarthy JS, Griffin PM, Sekuloski S, Bright AT, Rockett R, Looke D, Elliott S, Whiley D, Sloots T, Winzeler EA, Trenholme KR. Experimentally induced blood-stage Plasmodium vivax infection in healthy volunteers. J Infect Dis. 2013 Nov 15;208(10):1688-94. doi: 10.1093/infdis/jit394. Epub 2013 Aug 1. PMID 23908484
- [Background] Collins KA, Wang CY, Adams M, Mitchell H, Robinson GJ, Rampton M, Elliott S, Odedra A, Khoury D, Ballard E, Shelper TB, Lucantoni L, Avery VM, Chalon S, Moehrle JJ, McCarthy JS. A Plasmodium vivax experimental human infection model for evaluating efficacy of interventions. J Clin Invest. 2020 Jun 1;130(6):2920-2927. doi: 10.1172/JCI134923. PMID 32045385
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000212-I.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Malaria-naive US Adults Between 18 and 50 Years of Age: A single dose of cryopreserved inoculum containing blood-stage P. vivax will be administered IV
  HMPBS02-Pv: The blood-stage P. vivax master cell bank HMPBS02-Pv was also produced using blood collected from a consenting patient with naturally acquired malaria infection. The malaria infection was confirmed to be P. vivax by species-specific PCR at Pathology Queensland (accredited by the Australian National Association of Testing Authorities) and further confirmed by deep sequencing at the Sanger Institute. The clinical response to antimalarial chemotherapy was also demonstrated with this donor, who was successfully cured with artemether/lumefantrine.
Period: Overall Study
Arm/Group | Healthy Malaria-naive US Adults Between 18 and 50 Years of Age
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Malaria-naive US Adults Between 18 and 50 Years of Age
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  23 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: P. Vivax Blood Collection
Description: Collection of blood for the production of a P. vivax blood-stage parasite bank from study participants following experimental infection with P. vivax isolate HMPBS02-Pv.
Time Frame: Time of enrollment until blood collection for blood-stage parasite bank (10-11 days post-infection)
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Malaria-naive US Adults Between 18 and 50 Years of Age
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Time of enrollment until initiation of antimalarial treatment (10-11 days).
Arm/Group | Healthy Malaria-naive US Adults Between 18 and 50 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Malaria-naive US Adults Between 18 and 50 Years of Age (N=2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Chest discomfort (General disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Fatigue (General disorders) | 2 (4)
Haemoglobin decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (6)
Malaise (General disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (2)
Pyrexia (General disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT05095272/Prot_SAP_000.pdf